CLINICAL TRIAL: NCT07397845
Title: Stents Versus PAclitaxel Coated Balloons for Revascularization of CompleX and Small Coronary Vessels (SPARX) Trial
Acronym: SPARX RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Translumina GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TL/RCT/DEB/2025-04
Record Dates: First submitted 2026-01-05; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Drug Eluting Balloon; Drug Eluting Stent
Keywords: SPARX RCT; Protege
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, multi-centre, global, open label, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paclitaxel coated balloon (Experimental): Patients are only randomized after successful lesion preparations performed as per the the 3rd DCB Consensus. Post this, if the automatic generation of the device reflects Protege on the opted platform, then the patient is enrolled in this arm of the RCT
  Interventions: Device: Protégé and Protégé NC
- Drug coated balloon (Active Comparator): Patients are only randomized after successful lesion preparations performed as per the the 3rd DCB Consensus. Post this, if the automatic generation of the device reflects Agent on the opted platform, then the patient is enrolled in this arm of the RCT
  Interventions: Device: Agent
- Drug eluting stent (DES) (Active Comparator): DES to standard of care treatment during percutaneous coronary intervention. In this RCT, patients are only randomized after successful lesion preparations performed as per the the 3rd DCB Consensus. Post this, if the automatic generation of the device reflects DES (CE/FDA marked) on the opted platform, then the patient is enrolled in this arm of the RCT
  Interventions: Device: Drug Eluting Stent

INTERVENTIONS:
Device: Protégé and Protégé NC — Protégé Drug-eluting PTCA Balloon Catheters are rapid exchange catheters with a semi-compliant (Protégé DEB) balloon, or a non-compliant (NC) balloon (Protégé NC DEB), both with paclitaxel coating. Protégé is certified and CE marked.
  Arms: Paclitaxel coated balloon
Device: Agent — The AgentTM Paclitaxel-Coated Balloon Catheter (AgentTM DCB) is a monorail, semi-compliant PCI catheter. Agent™ PCB is CE and FDA certified and approved for clinical use both in Europe and in the US.
  Arms: Drug coated balloon
Device: Drug Eluting Stent — Drug Eluting stents is a standard of care treatment for narrowed coronary arteries of the patients
  Arms: Drug eluting stent (DES)

SUMMARY:
The main objective of the SPARX trial is to compare paclitaxel-coated balloons to with contemporary DES in complex and small coronary artery lesions in patients with NSTEACS or CCS; the co-primary objective is to compare two different paclitaxel-coated balloons, Protégé and Agent, with each other.

DETAILED DESCRIPTION:
PCI with DES remains a cornerstone of interventional cardiology for the treatment of coronary artery disease. While DES have significantly improved outcomes compared to plain old angioplasty (POBA) and metal stents, there is still a risk of in-stent restenosis (ISR) and stent thrombosis (ST). To overcome these problems, non-stent techniques using only DCBs have emerged as a way of delivering anti-proliferative drugs to the vessel wall without the need for a permanent implant. It is hypothesised that this approach may promote positive remodelling and reduce the risk of vessel thrombosis and restenosis.

The use of PCI with DCB alone was first investigated for the treatment of ISR, where it showed good results and is currently recommended in guidelines for the treatment of ISR. There have also been several DCB trials in de novo coronary lesions, but the results have been more mixed. Many DCBs are now commercially available, both with paclitaxel and sirolimus coating, and it appears that there is no "class effect" due to the heterogeneity that exists within balloon designs, polymer coating, type of drug and concentrations used.

One of the first trials in de novo lesions, the PICCOLETO trial, was stopped early due to a higher MACE rate in the DCB group compared to the DES group. However, several weaknesses of the study may explain the worse outcome in those treated with DCBs compared to DES. The most important was probably the low dose of paclitaxel delivered by the balloon and the fact that only a small percentage of the population underwent lesion predilatation. Several studies have later shown non-inferiority of DCB to DES for de novo lesions, and the method is currently embraced by the interventional cardiology community.

Several DCBs are now available and approved for use, and more are on the way, but head-to-head data are scarce. The SPARX trial is designed to compare two DCBs, Protégé™ and Agent™, with conventional DES PCI in complex and small coronary lesions, with the idea that this type of coronary disease may benefit from a DCB-only technique. The trial will also compare the two certified and well-established paclitaxel-coated balloons, Protégé™ and Agent™. The hypothesis is that Protégé™ will perform at least as well as Agent™.

The primary objective of the SPARX trial is to compare paclitaxel-coated balloons with contemporary DES in complex and small coronary artery lesions in patients with non-ST elevation acute coronary syndrome (NSTEACS) or chronic coronary syndrome (CCS); The co-primary objective is to compare 2 different paclitaxel-coated balloons, Protégé™ and Agent™, with each other.

ELIGIBILITY:
Clinical inclusion criteria:

1. Age≥18 years
2. Patient with NSTE-ACS or CCS with either symptoms and/or ischemia on non-invasive or invasive testing (i.e. FFR/iFR, CMR, SPECT, PET-CT or stress-echo)
3. The patient must be able to understand and provide written informed consent and comply with all study procedures
4. Life expectancy of > 2 years

   Angiographic inclusion criteria:
5. One or more trial target vessel (LAD, CX or RCA, or of their branches) with:

   1. Stenosis of ≥70% or
   2. Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia by positive stress test, or FFR ≤0.80, or iFR <0.90 or IVUS minimum lumen area ≤4.0 mm2
6. The target vessel/target lesion matches at least one of the following criteria

   1. Small vessel: vessel reference diameter is ≤ 3 mm
   2. Long lesions: length ≥ 25 mm
   3. Calcified lesion: grade 3 by angiography or confirmed on intravascular imaging
   4. Chronic total occlusion (CTO)
   5. Bifurcation lesions, including ostial LAD and ostial CX
   6. Lesions in diabetic coronary artery disease
   7. In-Stent Restenosis (ISR)
7. Lesion preparation must be according to the 3rd DCB consensus, with lesions that have:

   1. ≤ 30% residual stenosis
   2. TIMI (Thrombolysis in Myocardial Infarction) flow grade 3.
   3. The absence of flow-limiting dissection (Type A-C allowed only)

Clinical exclusion criteria:

1. STEMI or cardiogenic shock related to an acute MI within 2 days prior to the index PCI
2. Pregnancy or nursing declarations (As per country specific guideline) (a negative pregnancy test is required of women with child-bearing potential within 7 days prior to enrollment)
3. LVEF<30%
4. Known contraindication or hypersensitivity to any limus family drugs, paclitaxel, or to medications such as heparin, aspirin, clopidogrel, ticlopidine, prasugrel and ticagrelor or any component of the devices.
5. Allergy to imaging contrast media which cannot be adequately pre-medicated
6. Stroke/TIA during the last 6 months, or any prior intracranial hemorrhage
7. Active peptic ulcer or upper gastrointestinal bleeding within last 6 months
8. Known renal insufficiency with an eGFR<30 ml/min1.73m2, or subject on dialysis, or acute renal failure (as per physician judgment)
9. Planned surgery within 6 months with the necessity to stop DAPT
10. History of bleeding diathesis or coagulopathy
11. Platelet count<100.000 cells/mm3 or >400.000 cells/mm3, a WBC of <3000 cells/mm3, documented or suspected liver disease (including laboratory evidence of hepatitis)
12. Patient is a recipient of a heart transplant
13. Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation

    Angiographic exclusion criteria:
14. Target lesion is in the left main coronary artery
15. Target lesion is in a coronary artery bypass graft
16. Flow limiting target vessel thrombus
17. Evidence of aneurysm in target vessel within 10 mm of the target lesion
18. Aorto-ostial target lesion (within 3 mm of the aorta junction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Device oriented composite endpoint (DOCE) | 24 months
  1. Cardiac death
  2. New target vessel - related myocardial infarction (TV-MI)
  3. Ischemia-driven target-lesion revascularization (TLR)

SECONDARY OUTCOMES:
Patient oriented composite endpoint (POCE) | 1 month, 6 month, 12 month, 18 month, 24 month
  1. All-cause death
  2. Any Stroke
  3. All new MI (TV and non-TV related)
  4. Unplanned ischemia-driven repeat revascularization
Additional outcomes | 1 month, 6 month, 12 month, 18 month, 24 months
  Total no of events in 1380 patients will be analysed-
  1. Definite or probable vessel (stent) thrombosis
  2. Ischemia-driven target-vessel revascularization (TVR)
  3. Major bleeding (BARC type 3 to 5)

OTHER OUTCOMES:
All individual components of DOCE and POCE | 1 month, 6 month, 12 month, 18 month, 24 month
  Total no of events in 1380 patients will be analysed -
  1. All-cause death
  2. Cardiac death
  3. Any Stroke
  4. All new MI (TV and non-TV related)
  5. Ischemia-driven TLR
  6. Unplanned ischemia-driven repeat revascularization
Other outcomes of interest | 0 day (during index PCI)
  Device success: Defined as the ability of the study devices to be delivered, dilated and retrieved from the target lesion during index procedure.
Other outcomes of interest | 0 day (during index PCI)
  Procedure duration, radiation exposure and contrast volume.
Other outcomes of interest | 7 days
  Procedural success: Achievement of a final diameter stenosis of < 30% (site-reported) using any PCI method, without the occurrence of death, MI or repeat vessel revascularization during index- hospital stay.
Other outcomes of interest | 7 days
  Acute or subacute vessel closure/thrombosis: diameter stenosis of 100% and/or TIMI flow grade 0.
Other outcomes of interest | 2 days
  Periprocedural myocardial injury within 48 hours (according to SCAI definition): Elevated CK-MB of >10 times upper limit of normal, or cTn (T or I)>70 times upper limit of normal within 48 hours from the procedure. If cardiac biomarker levels are elevated before the procedure, these levels will be used as the reference instead of normal values.
Other outcomes of interest | 7 days
  Length of In-hospital stay (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Florim Cuculi, MD, Principal Investigator — Cardiology Division Heart Center - Luzerner Kantonsspital Spitalstrasse, 6000 Luzern 16, Switzerland; Prof. Dr. Adnan Kastrati, MD PhD, Study Chair — German Heart Center Munich Lazarettstraße 36, 80636 München, Germany

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share individual participant data. However, an overall study data and it's publication results shall be uploaded upon completion of this project at Ct.Gov.